CLINICAL TRIAL: NCT02376452
Title: Phase II Study of 2-weekly Raltitrexed Plus Irinotecan Regimen (RAILIRI) Versus Fluorouracil, Leucovorin, and Irinotecan Regimen (FOLFIRI) as Second-line Treatment in Advanced Colorectal Cancer Patients
Brief Title: Phase II Study of 2-weekly RAILIRI Versus FOLFIRI as Second-line Treatment in Advanced Colorectal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jin Li, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RALIRI
Record Dates: First submitted 2015-02-12; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — raltitrexed; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RALIRI (Experimental): Raltitrexed combined with irinotecan
  Interventions: Drug: Raltitrexed; Drug: Irinotecan
- FOLFIRI (Placebo Comparator): 5-fluorouracil,folinate combined with irinotecan
  Interventions: Drug: Irinotecan; Drug: 5-fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Raltitrexed — 2mg/m2 iv gtt, d1
  Arms: RALIRI
Drug: Irinotecan — 180 mg/m2 iv gtt, d1
Drug: 5-fluorouracil — 5-FU 400mg/m2 iv, 2400mg/m2 civ 46h
  Other Names: 5-FU
  Arms: FOLFIRI
Drug: Leucovorin — 400mg/m2 iv gtt,d1
  Other Names: LV
  Arms: FOLFIRI

SUMMARY:
This study is designed to compare the efficacy and safety of two-weekly RAILIRI regimen with FOLFIRI regimen in the treatment of advanced colorectal cancer patients in the second-line setting.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years with histologically or cytologically confirmed advanced colorectal adenocarcinoma
* Eastern Cooperative Oncology Group performance status of 0 to 1
* life expectancy of ≥ 3 months
* patients who had failed first-line treatment with either XELOX (capecitabine combined with oxaliplatin) or FOLFOX (5-fluorouracil/leucovorin with oxaliplatin)
* at least one measurable disease lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria
* have adequate bone marrow, hepatic, and renal function

Exclusion Criteria:

* patients with previous chronic inflammatory bowel disease, chronic diarrhea or recurrent bowel obstruction
* patients with symptomatic brain metastases
* active clinical severe infection
* previously received irinotecan or raltitrexed
* dihydropyrimidine dehydrogenase (DPD) enzyme adequate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2 months

SECONDARY OUTCOMES:
overall survival | 6 months
overall response rate | 2 months
disease control rate | 2 months
Number of Participants with Adverse Events | 2 months
quality of life questionnaire | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, Principal Investigator — Medical Oncology, Fudan University Shanghai Cancer Center
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China